CLINICAL TRIAL: NCT01399268
Title: Effect of Steroids Given Over 24 Hours on Cytokine Release and Urinary Desmosine Levels in Patients Undergoing Bilateral Total Knee Replacement
Brief Title: Steroids in Bilateral Total Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSS-28116
Record Dates: First submitted 2011-07-14; First posted 2011-07-21 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Postoperative Inflammatory Response
Keywords: Bilateral total knee replacement; cytokine; desmosine
MeSH Terms: interventions — Hydrocortisone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Steroid (Experimental): Hydrocortisone 100 mg IV Q 8hrs x3
  Interventions: Drug: Hydrocortisone
- Control (Placebo Comparator): Saline IV Q8hr x3
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Hydrocortisone — Prepared by pharmacy, 100 mg, IV, every 8 hours, 3 times
  Arms: Steroid
Drug: Saline — Prepared by pharmacy same volume as study drug, IV, every 8 hours 3 times
  Arms: Control

SUMMARY:
Inflammation related to cytokine release is known to occur with surgery. The cytokine IL6, a major marker of inflammation is known to increase during total joint replacement surgery. IL6 has been found to be elevated postoperatively in patients with hip fractures and has been linked to mental status changes and possibly other complications. It is known to lead to shock and participate in the inflammatory state seen in sepsis. High levels have further been linked to postoperative fever, confusion, symptoms of depression, acute respiratory distress syndrome (ARDS) and fat embolism syndrome (FES). Previously the investigators found that low dose steroids given in two doses in the initial perioperative period decreased the amount of IL6 released compared to placebo, but this was not sustained past 24 hours.

Desmosine is a stable breakdown product of elastin from lung tissue that can be measured in urine samples. It is considered to be a marker of lung injury and is found to be elevated in patients with ARDS, congestive obstructive pulmonary disease and FES. Previously, the investigators have found that urine desmosine levels rise with bilateral total knee replacement compared to unilateral total knee replacement indicating possible lung injury.

Therefore the investigators hypothesize:

Continued low dose steroids given three times over a 24 hour period will:

1. Significantly decrease peak IL6 cytokine release during bilateral total knee replacement and maintaining this reduction in IL6 beyond 24 hours.
2. Decrease urinary desmosine levels, and hence be protective of lung injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for bilateral total knee replacement
* Between 50-90 years of age

Exclusion Criteria:

* Patients on steroid therapy
* Patients that require stress-dose steroid pre-operatively
* Patients that smoke
* Patients that are diabetic
* Patients younger than 50 or older than 90 years

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2010-08 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kethy Jules-Elysee, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Derived] McLawhorn AS, Poultsides LA, Sakellariou VI, Kunze KN, Fields KG, Jules-Elysee K, Sculco TP. Low-Dose Perioperative Corticosteroids Can Be Administered Without Additional Morbidity in Patients Undergoing Bilateral Total Knee Replacement: A Retrospective Follow-up Study of a Randomized Controlled Trial. HSS J. 2022 Feb;18(1):48-56. doi: 10.1177/15563316211006098. Epub 2021 Apr 9. PMID 35087332

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Steroid | Control
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Steroid | Control | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (7) | 71 (9) | 67.5 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 6 | 9 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Decrease in IL6 Level
Time Frame: 24 hours postoperative
Measure: Mean (99% Confidence Interval); unit: pg/ml
Arm/Group | Steroid | Control
Number analyzed (Participants) | 15 | 15
pg/ml | 359.4 [300 to 400] | 381.6 [300 to 400]

2. Secondary Outcome: Desmosine Level
Time Frame: 24 hours postoperative
Population: Data were not collected
Arm/Group | Steroid | Control
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

3. Secondary Outcome: Blood Glucose
Time Frame: 24 hours postoperative
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Steroid | Control
Number analyzed (Participants) | 15 | 15
mg/dL | 133 (30) | 102 (17)

4. Secondary Outcome: Length of Hospital Stay
Time Frame: Length of hospital stay, an expected average of 5 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Steroid | Control
Number analyzed (Participants) | 15 | 15
days | 5 (0.9) | 5 (0.8)

5. Secondary Outcome: In Hospital Infection Rate
Time Frame: Length of hospital stay, an expected average of 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid | Control
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

6. Secondary Outcome: Mortality
Time Frame: Length of hospital stay, an expected average of 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid | Control
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

7. Secondary Outcome: Ability to Ambulate
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid | Control
Number analyzed (Participants) | 15 | 15
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: The study collected data for 30 days after surgery
Arm/Group | Steroid | Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes